CLINICAL TRIAL: NCT03484481
Title: Positive Incomes of Nutritional Support Modalities in Terms of Nutritional Status and Inflammation in Hemodialysis Patients With Severe Malnutrition
Brief Title: Incomes of Nutritional Support Modalities in Hemodialysis Patients With Severe Malnutrition
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Bahar Gurlek Demirci, MD, Baskent University
Other Study IDs: 3558238bc
Record Dates: First submitted 2018-03-24; First posted 2018-03-30 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Severe Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1;Oral nutritional support (ONS): patients ongoing hemodialysis who received only oral nutritional support (Nutrena) and refused intradialytic parenteral nutrition; n: 14
  Interventions: Dietary Supplement: Oral Nutritional Support; Nutrena
- 2; Intradialytic Parenteral Nutrition: patients ongoing hemodialysis who received only Intradialytic Parenteral Nutrition (Kabiven central) and refused parenteral nutrition; n: 14
- group 3; combination group: patients ongoing hemodialysis received both ONS and Intradialytic Parenteral Nutrition NS; n: 10
  Interventions: Dietary Supplement: Oral Nutritional Support; Nutrena; Dietary Supplement: Intradialytic Parenteral Nutrition; Kabiven central
- group 4; dietetic support group;: patients ongoing hemodialysis who refused all types of nutritional support and only followed by counselling, n: 18

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Support; Nutrena — Patients in group 1 and 3 take ONS 200 ml/day twice a day at home. Patients in group 2 and 3 received IDPN administrations. ]. Its infusion was started 30 minutes after initiation of HD via the venous port of the bubble trap on the HD tubing and continued throughout the entire HD procedure at a rate of 150 ml/h for 30 min and consisted of 300 ml for 3 hour.
  Groups: 1;Oral nutritional support (ONS); group 3; combination group
Dietary Supplement: Intradialytic Parenteral Nutrition; Kabiven central — Patients in group 2 and 3 received IDPN administrations Its infusion was started 30 minutes after initiation of HD via the venous port of the bubble trap on the HD tubing and continued throughout the entire HD procedure at a rate of 150 ml/h for 30 min and consisted of 300 ml for 3 hour.
  Groups: group 3; combination group

SUMMARY:
Introduction: Protein energy malnutrition is one of the strongest predictors of morbidity and mortality in maintenance hemodialysis (MHD) patients. Many reports indicate that there is a high prevalence of malnutrition up to 40% , and has a strong association with inflammation and cardiovascular disease (CVD) as well as lower quality of life in this population. The aim of this study was to compare the nutritional modalities by means of biochemical parameters, arterial stiffness and bioimpedance analysis.

Material and Methods: We designed an observational study with 56 malnourished MHD patients (mean age: 61.8±12.3 years, duration of hemodialysis: 7.9±5.1 years) . Patients were distributed into 4 groups according to patients requests for nutritional support modalities. We offered the combination of oral nutritional support (ONS) and intradialytic parenteral nutrition (IDPN) to all patients however some of the patients refused this combination thus we had 4 groups as; Group 1 (patients received only ONS and refused parenteral nutrition; n: 14), group 2 (patients received only parenteral NS and refused ONS; n: 14), group 3 (patients received both oral and parenteral NS; n: 10) and group 4 (dietetic support group; patients who refused all types of nutritional support and only followed by counselling, n: 18) for 12 months. Biochemical parameters were assessed from monthly clinical visits. Normalized protein catabolic rate (nPCR), malnutrition-inflammation score (MIS), body composition (fat mass [FM], fat-free mass (FFM) muscle mass (MM, body mass index (BMI)) by multifrequency bioimpedance analysis (BCM, Fresenius).

DETAILED DESCRIPTION:
Our current standard nutrition care is based upon existing recommendations and involves nutrition counselling for optimal dietary intake from food and beverages, food fortification, administration of oral nutrition supplementation (ONS) and/or IDPN in malnourished MHD patients.

Among 712 MHD patients, 138 who were diagnosed as severely malnourished (subjective global assessment (SGA) scores are B/C and serum albumin concentration <3.5 g/dL and/or a loss of ≥5% dry weight (DW) over the past 3 months ) were followed up between January 2016 - December 2016.

The patients whose at least 6 months interrupted data could be obtained under the recomemded nutritional support were included. Exclusion criteria were as follows; active infectious disease, chronic inﬂammatory systemic diseases (CIDs) like rheumatoid arthritis, systemic lupus erythematosus and multiple sclerosis, malabsorption syndrome, those treated with steroids or antiandrogens, inadequate dialysis (single pool Kt/V < 1.4), recent surgery within 3 months or during follow-up; hospitalization at time of randomization; nephrotic syndrome; active malignancy or history of malignancy.

eigthy-two patients were excluded according to above criteria thus 56 severely malnourished patients data was included to the study and are recommended to receive ONS and/or IDPN. The given supplementation is continued until the nutritional parameters are ameliorated. The patients choice was the determinator of the received nutritional support.

Patients were distributed into 4 groups according to patients requests for nutritional support modalities. We offered the combination of ONS and IDPN to all patients however some of the patients refused this combination thus we had 4 groups as; Group 1 (patients received only ONS and refused parenteral nutrition; n: 14), group 2 (patients received only parenteral NS and refused ONS; n: 14), group 3 (patients received both oral and parenteral NS; n: 10) and group 4 (dietetic support group; patients who refused all types of nutritional support and only followed by counselling, n: 18) (Figure 1: Study Flowchart).

All patients gave informed consent for this study, which was approved by the ethics committee of Baskent University School of Medicine.

Nutritional supplementation Each patient was consulted monthly by a dietitian to achieve the target calorie intake of 35 kcal/kg/day. A snack providing approximately 300 kcal, 14 g protein, 55 g carbohydrate, and 10 g fat was served to all patients during the sessions.

- Oral Nutrition Support (ONS): Patients in group 1 and 3 take ONS 200 ml/day twice a day at home. Each serving (200 mL) of ONS preparation (Nutrena;Abbott Nutrition, Zwolle, Holland) contained 400 kcal, 14 g protein, 41.3 g carbohydrate, and 19.2 g fat and had lower concentrations of sodium, potassium, and phosphorus than standard ONS. ONS consumption was recorded at each dialysis session.

- Intradialytic Parenteral Nutrition (IDPN) Patients in group 2 and 3 received IDPN administrations [(Kabiven central; a sterile, hypertonic emulsion, for central venous administration, in a Three Chamber Bag; the solution contains dextrose solution for fluid replenishment and caloric supply amino acid solution with electrolytes, which comprises essential and nonessential amino acids provided with electrolytes and Intralipid® 20% (a 20% Lipid Injectable Emulsion), prepared for intravenous administration as a source of calories and essential fatty acids]. Its infusion was started 30 minutes after initiation of HD via the venous port of the bubble trap on the HD tubing and continued throughout the entire HD procedure at a rate of 150 ml/h for 30 min and consisted of 300 ml for 3 hour.

ELIGIBILITY:
Inclusion Criteria:

* subjective global assessment (SGA) scores B or C
* serum albumin concentration <3.5 g/dL
* loss of ≥5% dry weight (DW) over the past 3 months )

Exclusion Criteria

* active infectious disease,
* chronic inﬂammatory systemic diseases (CIDs) like rheumatoid arthritis, systemic lupus erythematosus
* multiple sclerosis
* malabsorption syndrome
* inadequate dialysis (single pool Kt/V < 1.4)
* recent surgery within 3 months or during follow-up;
* hospitalization at time of randomization
* nephrotic syndrome
* active malignancy or history of malignancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among 712 MHD patients, 138 who were diagnosed as severely malnourished were followed up between January 2016 - December 2016. Eigthy-two patients were excluded according to above criteria thus 56 severely malnourished patients data was included to the study and are recomended to receive ONS and/or IDPN. The given supplementation is continued until the nutritional parameters are ameliorated. The patients choice was the determinator of the received nutritional support.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Inflammation | 12 months
  C-reactive protein